CLINICAL TRIAL: NCT04090242
Title: An Assessment of the Impact of an App Based Diabetes Training Program in Conjunction With the Use of BD Nano 2nd Gen 4mm Pen Needle on Diabetes Self-efficacy in People With Type 2 Diabetes
Brief Title: Impact of App Based Diabetes Training Program in Conjunction With the BD Nano Pen Needle in People With T2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment halted prematurely due to the Covid-19 pandemic
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DBC-19BRGHT02
Record Dates: First submitted 2019-08-28; First posted 2019-09-16 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- App plus Nano (Active Comparator): Use of BD Diabetes Care Application for Mobile devices PLUS the use of BD Nano 2nd Gen Pen Needle for delivery of insulin
  Interventions: Device: BD Diabetes Care Application (for mobile devices) PLUS use of BD Nano Pen Needle
- Standard Care (No Intervention): Standard of Care/Subject is to continue on their current diabetes management regime

INTERVENTIONS:
Device: BD Diabetes Care Application (for mobile devices) PLUS use of BD Nano Pen Needle — Subjects in the Intervention Group will be instructed to use the DC-App and switch from their current pen needle to the BD Nano 2nd Gen Pen needle during their participation in the study. The app is intended to be used as a patient education tool and data logger to augment the diabetes care team.
  Arms: App plus Nano

SUMMARY:
This is a multi-center, open-label, parallel-group, randomized controlled study in subjects with type 2 diabetes using multiple daily injection (MDI) insulin therapy. Subjects will be randomized to either receive the DC App and BD Nano 2nd Gen pen needles (intervention) or continue their standard of care using their current pen needle and diabetes management (control). The study will consist of four visits and two scheduled phone calls across a total of 10 weeks.

DETAILED DESCRIPTION:
At Visit 1 (Day -14) site staff will screen and enroll qualified subjects, provide a BGM (Accu-Chek Guide) and attach a blinded flash glucose sensor (Libre Freestyle) to the back of the arm. Subjects will complete any applicable baseline Patient Reported Outcomes (PRO) questionnaires and be sent home with no changes to their current therapy. While at home Subjects will be asked to test blood glucoses using the provided BGM and continue their usual insulin dosing before returning to clinic for Visit 2. Visit 2 will consist of randomization (Interventional Group or Control Group). The control group will be continued on their current pen needle and receive standard visit education as needed. The intervention group will be trained on the use of the DC App and be switched to BD Nano 2nd Gen pen needle. During weeks 3 through 8, subjects in both groups will continue their usual insulin routine, with the control group adhering to their usual practice of managing their diabetes and the intervention group utilizing the DC app for relevant educational content and tips plus using the BD Nano 2nd Gen for all insulin injections. During Visit 3 subjects will get a 2nd fGM sensor placed and be instructed to continue their insulin routine for the final 2 weeks. Visit 4 is the last visit where subjects will have their fGM removed, return the BGM, complete applicable PRO surveys, an injection technique questionnaire and be discharged.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age minimum
2. Adult subjects with type 2 diabetes mellitus on Multiple daily injections (MDI) and giving themselves at least 2 injections of insulin / day using a pen injector. This may include at minimum i. giving 1 basal injection and at least 1 meal time injection or ii. giving at least 2 daily injections of mixed insulins or iii. giving 2 meal time injections iv. two injections of basal insulin per day will not be considered MDI for this study v. additional OAD/non-insulin injectable therapy is acceptable
3. Must currently be on MDI insulin therapy for at least 6 months prior to enrollment and, in the opinion of the investigator, would benefit from dose optimization.
4. Willing to use the BD provided BGM for the study duration.
5. Hemoglobin A1C of 8.0 - 11% at screening (tested at enrollment unless Subject has a documented HbA1c value on file at the site that was drawn within 3 months of enrollment date).
6. In stable health status with no acute or significant illness, based on the opinion of the investigator.
7. Able to read, write and follow instructions in English (translations will not be provided).
8. Currently using a smartphone and able to understand the use of mobile apps.
9. Able and willing to provide informed consent.
10. Able and willing to follow study procedures.

Exclusion Criteria:

* Subjects with any one of the following characteristics will be excluded from participation:

  1. Pregnant or breast feeding- self reported.
  2. Subject on basal-only
  3. Uncontrolled comorbidities or acute illness
  4. Currently using Nano 2nd Gen pen needles
  5. Use of a smartphone with iOS 10.0 or lower or with Android OS 5.0 "Lollipop" or lower
  6. Use of CGM or fGM less than 6 months and not proficient in its use, however this may be left up to the investigators discretion.

     i. Subjects may continue to wear their own CGM/fGM during their participation in this study if they adhere to the testing of blood glucose using the site provided BGM.
  7. Subjects not on stable doses of concomitant non-insulin diabetes medications. Stable is defined as not requiring new non-insulin diabetes medications or any changes in dosing of current non-insulin diabetes medication during study participation (10 weeks) unless warranted by investigator for the safety of the subject.
  8. Actively using one of the following diabetes management apps deemed similar and not willing to stop using it during participation on the study (exclusionary apps; Onedrop, Welldoc (Bluestar), Dario, Sugar Sense Glucose, Buddy, mySugr, Omada, Livongo, Accu-Check Connect, SugarIQ).
  9. Known sensitivity to adhesives.
  10. Currently using the DC app.
  11. Employed by, or currently serving as a contractor or consultant to BD or study site
  12. Any other condition the investigator deems to pose a risk to the Subject in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Mahoney, PhD, Study Director — Becton Dickinson; David Klonoff, M.D, FACP, Principal Investigator — Diabetes Research Institute, Mills-Peninsula Medical Center, California
Locations (4):
- United States (4):
  - Mills Pennisula Medical Center-Diabetes Research Institute, San Mateo, California
  - Metabolic Research Institute, West Palm Beach, Florida
  - East West Medical Research Institute, Honolulu, Hawaii
  - Texas Diabetes and Endocrinology, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | App Plus Nano | Standard Care
Started | 28 | 30
Completed | 27 | 30
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | App Plus Nano | Standard Care | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.8) | 59.4 (10.8) | 58.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 9 | 18 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 21 | 26 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 16 | 33
  Asian | 6 | 6 | 12
  Black or African American | 3 | 5 | 8
  Other | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58
Current Use of Diabetes App [Count of Participants; unit: Participants]
  No | 26 | 29 | 55
  Yes | 2 | 1 | 3
Use of Continuous Blood Glucose Monitoring System [Count of Participants; unit: Participants]
  No | 16 | 19 | 35
  Yes | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Attitude Toward Diabetes - Diabetes Empowerment Scale (DES) From Baseline to End of Study
Description: A standardized questionnaire including 8 questions with response categories of 'strongly disagree', 'somewhat disagree', 'neutral', 'somewhat agree', and 'strongly agree'. An overall score for the DES is calculated by summing all of the item scores and dividing by 8 for a possible score range of 1-5 where a higher score indicates a higher level of empowerment.
Time Frame: Baseline (Day -14) and Study End (Day 56)
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Scores on scale
  Baseline | 4.16 (0.55) | 4.09 (0.66)
  End of Study | 4.17 (0.84) | 4.26 (0.52)
Statistical Analysis 1: Comparison: App Plus Nano vs Standard Care; With assumptions made in statistical analysis plan, a sample size of 43 subjects per arm had >80% power to detect a significant difference between the two arms (based on a 2-sided t-test, 95% CI for DES difference between groups). Adding a 10% buffer, planned enrollment was 96 subjects. However, enrollment ended early with about 25 subjects in each arm (56 subjects total). Thus, power decreased to 56%. The study was not sufficiently powered under these conditions; Test type: Other; p = 0.392, Mixed Models Analysis — The p value is for the comparison between interventional and control group on change of DES score between baseline and end of study; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.53 to 0.21]

2. Secondary Outcome: Change in 24 Hour Average Blood Glucose From Baseline to End of Study
Description: Freestyle Libre Pro blinded flash glucose monitoring will be used to assess change in average 24 hour blood glucose between groups Subjects will wear Libre sensors on the backs of their arm for the 2 weeks at the beginning of the study and 2 weeks at the end of the study.
Time Frame: Baseline (Day -14 through Day -1) and Study End (Day 42 through Day 56)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
mg/dl
  Baseline | 187.0 (39.7) | 161.8 (37.9)
  End of study | 184.9 (55.7) | 173.1 (45.3)

3. Secondary Outcome: Blood Glucose Values in Range of <54 mg/dL at Baseline Compared to End of Study
Description: Data collected by the flash glucose monitor were used to calculate percent of time in range to compare differences between groups at baseline and study end. For example, Time below 54 mg/dl is calculated in the following manner: Number of all glucose data points below 54 mg/dl / total number of glucose data points X 100. Since data points are all 5 minutes apart, this calculation provides the percentage of time in that range.
Time Frame: Baseline (Day -14 through Day -1) and Study End (Day 42-through Day 56)
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Percent of time
  Baseline | 0.73 (1.11) | 2.68 (5.14)
  End of study | 0.83 (1.05) | 1.07 (1.25)

4. Secondary Outcome: Blood Glucose Values in Range of <70 mg/dL at Baseline Compared to End of Study
Description: Data collected by the flash glucose monitor were used to calculate percent of time in range to compare differences between groups at baseline and study end.
Time Frame: Baseline (Day -14 through Day -1) and Study End (Day 42-through Day 56)
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Percent of time
  Baseline | 2.54 (3.18) | 6.37 (9.31)
  End of study | 3.34 (3.46) | 3.46 (3.46)

5. Secondary Outcome: Blood Glucose Values Between 70 mg/dL and 180 mg/dL at Baseline Compared to End of Study
Description: as for outcome 4
Time Frame: Baseline (Day -14 through Day -1) and Study End (Day 42-through Day 56)
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Percent of time
  Baseline | 49.35 (18.93) | 58.75 (18.58)
  End of study | 51.85 (23.17) | 57.19 (23.43)

6. Secondary Outcome: Blood Glucose Values in Range of >180mg/dL at Baseline Compared to End of Study
Description: as for outcome 4
Time Frame: Baseline (Day -14 through Day -1) and Study End (Day 42-through Day 56)
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Percent of time
  Baseline | 48.11 (20.20) | 34.88 (22.0)
  End of study | 44.82 (24.79) | 39.35 (24.82)

7. Secondary Outcome: Blood Glucose Values in Range of >250 mg/dL at Baseline Compared to End of Study
Description: as for outcome 4
Time Frame: Baseline (Day -14 through Day -1) and Study End (Day 42-through Day 56)
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Percent of time
  Baseline | 18.92 (17.67) | 11.29 (11.11)
  End of study | 19.29 (21.09) | 15.54 (18.49)

8. Secondary Outcome: Change in Mean Amplitude of Glycemic Excursion (MAGE) Between Baseline and End of Study
Description: Flash glucose monitoring data were used to measure glycemic variability changes at baseline and study end between groups. Measuring glycemic variability helps determine how much glucose levels change over the course of a day or between days.
Time Frame: Baseline (Day -14 through Day -1) and Study End (Day 42 through Day 56)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
mg/dl
  Baseline | 133.64 (26.38) | 121.68 (19.99)
  End of study | 127.57 (25.04) | 124.16 (19.12)

9. Secondary Outcome: Change in Diabetes Distress Screening Scale - 17 (DDS17) Scores From Baseline to End of Study
Description: A standardized questionnaire including 17, 6-point Likert Scale questions where 1 indicates "Not a problem", 2 indicates "A slight problem", 3 means "A moderate problem", 4 indicates a "Somewhat serious problem", 5 indicates "A serious problem", and 6 means "A very serious problem". Using this scale, a Total Score, Emotional Burden Score, Physician Score, Regimen Distress Score, and Interpersonal Score were calculated.
Time Frame: Baseline (Day -14) to Study End (Day 56)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Score on a scale
  Total Score (Baseline) | 1.81 (0.66) | 2.03 (0.92)
  Total Score (End of Study) | 1.83 (0.61) | 2.10 (1.01)
  Emotional Burden Subscale (Baseline) | 2.19 (1.22) | 2.19 (1.08)
  Emotional Burden Subscale (End of Study) | 2.21 (1.06) | 2.17 (1.09)
  Physician Distress Subscale (Baseline) | 1.01 (0.05) | 1.48 (1.10)
  Physician Distress Subscale (End of Study) | 1.05 (0.20) | 1.48 (1.14)
  Regimen Distress Subscale (Baseline) | 2.23 (0.86) | 2.39 (1.10)
  Regimen Distress Subscale (End of Study) | 2.16 (0.73) | 2.43 (1.07)
  Interpersonal Distress Subscale (Baseline) | 1.57 (0.90) | 1.89 (0.98)
  Interpersonal Distress Subscale (End of Study) | 1.69 (1.05) | 2.24 (1.35)

10. Secondary Outcome: Insulin Delivery System Rating Questionnaire (IDSRQ) Scores at Baseline and End of Study
Description: A standardized questionnaire including several questions with ordinal response scales from 1 to 4 and 1 to 5. The IDSRQ has seven sub-scales (satisfaction, interference of treatment with daily activities, diabetes-related worries, clinical efficacy, psychological well-being, social burden, and treatment preference). Each sub-scale is calculated as a mean of their corresponding items with scores ranging from 0-100. Higher scores represent higher levels of satisfaction, perceived clinical efficacy, and psychological well-being, interference with daily activities, diabetes-related worries, and social burden.
Time Frame: Baseline (Day -14) and Study End (Day 56)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
Score on a scale
  Satisfaction Subscale (Baseline) | 67.83 (2.45) | 66.45 (23.46)
  Satisfaction Subscale (End of Study) | 72.76 (22.20) | 69.72 (18.89)
  Interference Subscale (Baseline) | 25.31 (15.49) | 17.95 (20.57)
  Interference Subscale (End of Study) | 27.01 (19.85) | 25.28 (21.81)
  Clinical Efficacy Subscale (Baseline) | 58.02 (21.34) | 53.24 (21.48)
  Clinical Efficacy Subscale (End of Study) | 58.85 (22.03) | 53.70 (19.54)
  Diabetes-Related Worry Subscale (Baseline) | 41.98 (22.26) | 40.00 (18.30)
  Diabetes-Related Worry Subscale (End of Study) | 42.28 (23.48) | 39.31 (19.26)
  Social Burden Subscale (Baseline) | 35.19 (19.83) | 37.58 (16.36)
  Social Burden Subscale (End of Study) | 32.80 (16.28) | 35.12 (16.78)
  Well-Being Subscale (Baseline) | 42.28 (12.01) | 43.94 (13.24)
  Well-Being Subscale (End of Study) | 47.41 (13.49) | 44.33 (13.65)
  Treatment Preference Subscale (Baseline) | 64.20 (14.74) | 57.08 (15.29)
  Treatment Preference Subscale (End of Study) | 63.35 (13.66) | 59.31 (14.46)

11. Secondary Outcome: Adherence to Refills and Medications Scale for Diabetes (ARMS-D) Questionnaire Scores at Baseline and Study End
Description: A standardized questionnaire including 11 multiple choice questions. The ARMS-D yields a total score plus two sub-scale scores (refill sub-scale and medication taking sub-scale. Items 1-10 are scored as follows: 1= none of the time, 2 = some of the time, 3 = most of the time, and 4 = all of the time. Item 11 is reversed scored. The ARMS-D total is a sum of all items for a possible score ranging from 11-44. The ARMS-D refill sub-scale is a sum of 4 items for a possible score ranging from 4-16. The ARMS-D medication taking sub-scale is a sum of 7 items for a possible score ranging from 7-28. Lower scores indicate better adherence.
Time Frame: Baseline (Day -14) to Study End (Day 56)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 27 | 30
score on a scale
  ARMSD Total Score (Baseline) | 15.67 (3.46) | 16.57 (4.08)
  ARMSD Total Score (End of Study) | 16.07 (3.65) | 15.43 (3.07)
  Refill Subscale (Baseline) | 5.30 (1.51) | 6.07 (2.07)
  Refill Subscale (End of Study) | 5.37 (1.50) | 5.30 (1.37)
  Medication Taking Subscale (Baseline) | 10.37 (2.79) | 10.50 (2.54)
  Medication Taking Subscale (End of Study) | 10.70 (2.71) | 10.13 (2.42)

12. Secondary Outcome: Patient Satisfaction at Study End
Description: A questionnaire including 16, 5-point Likert Scale questions where 1 indicates strongly disagree and 5 indicates strongly agree. This questionnaire yields a total satisfaction score plus three sub-scale scores (mobile app satisfaction, pen needle satisfaction, and injection management system satisfaction). The total score ranges from 16-80. The mobile app and pen needle satisfaction sub-scale score range from 6-30 and is a sum of all items in the associated sub-scale. The management system sub-scale score ranges from 4-20 and is a sum of all items in the sub-scale. Higher scores indicate higher satisfaction.
Time Frame: Administered to participants in the Intervention group only at end of study (Day 56)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App Plus Nano
Number analyzed (Participants) | 27
score on a scale
  Patient Satisfaction Subscale | 63.52 (15.93)
  Mobile App Subscale | 21.96 (6.66)
  Pen Needle Subscale | 25.30 (6.35)
  System Subscale | 16.26 (4.38)

13. Other Pre Specified Outcome: Number of Hypoglycemic Events (<70mg/dL and <54mg/dL) at Baseline and Study End
Description: Frequency of hypoglycemia: The number of hypoglycemic events (<70mg/dL and <54mg/dL) as measured by blood glucose monitor (BGM) will be collected to determine frequency of hypoglycemia in each group.
Time Frame: Baseline (Day -14) to Study End (Day 56)
Measure: Mean (Standard Deviation); unit: Hypoglycemic events
Arm/Group | App Plus Nano | Standard Care
Number analyzed (Participants) | 28 | 30
Hypoglycemic events
  % time <54 mg/dL (Baseline) | 0.7 (1.1) | 2.7 (5.1)
  % time <54 mg/dL (Study End) | 0.8 (1.1) | 1.1 (1.3)
  % Time < 70 mg/dl (Baseline) | 2.5 (3.2) | 6.4 (9.3)
  % Time < 70 mg/dl (End of Study) | 3.3 (3.5) | 3.5 (3.5)

14. Other Pre Specified Outcome: Number of Hours of Patient Engagement With App
Description: Patient Engagement: Engagement with The DC App will be measured by app collected usage analytics and main assessment was time spent within app.
Time Frame: Baseline (Day 1) to Study End (Day 56)
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | App Plus Nano
Number analyzed (Participants) | 27
Hours | 7.2 (20.1)

ADVERSE EVENTS:
Time Frame: Adverse events reported between week 1 and week 10 of the study.
Arm/Group | App Plus Nano | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/30
Other Adverse Events (participants affected / at risk) | 2/27 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | App Plus Nano (N=27) | Standard Care (N=30)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | App Plus Nano (N=27) | Standard Care (N=30)
Upper respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Common Cold (General disorders) | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04090242/Prot_SAP_000.pdf